CLINICAL TRIAL: NCT04290923
Title: Determination of Blood Tumor Cells Using Magnetic Nanoparticles
Brief Title: Determination of Blood Tumor Cells
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01140
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Abnormalities Cell Epithelial
Keywords: Epithelial Cell Adhesion Molecule; Magnetite Nanoparticles; Tumor cells
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Colorectal Cancer, Hereditary Nonpolyposis, Type 8

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample at one single time point
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Magnetic nanoparticles coated with anti-EpCAM or anti-CD52 antibodies will be tested ex-vivo in patients blood .

DETAILED DESCRIPTION:
Magnetic nanoparticles, coated with epithelial cell adhesion molecule (EpCAM)-antibodies are designed to interact with epithelial tumor cells. Aim of this study is to see if circulating tumor cells (EpCAM as marker)can be removed out of the blood with the help of these particles. Patients suffering from prostate, colon, lung or pancreatic cancer will be asked to test their blood.

Similarly, magnetic nanoparticles will be coated with antibodies, directed against non-solid tumors in the blood such as lymphoma or leukemia (CD52 as marker).

ELIGIBILITY:
Inclusion Criteria:

Epithelial cell cancer, advanced stage Non-solid tumors (lymphoma, leukemia)

Exclusion Criteria:

Inability to understand the language of the center (German)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Criterion for the enrollment is the presence of an epithelial cell carcinoma or the presence of a non-solid tumor (i.e. lymphoma or leucemia)
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Number of CTC / lymphocytes removed | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice H Beck Schimmer, Prof, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Background] Herrmann IK, Bernabei RE, Urner M, Grass RN, Beck-Schimmer B, Stark WJ. Device for continuous extracorporeal blood purification using target-specific metal nanomagnets. Nephrol Dial Transplant. 2011 Sep;26(9):2948-54. doi: 10.1093/ndt/gfq846. Epub 2011 Feb 10. PMID 21310738
- [Background] Herrmann IK, Schlegel A, Graf R, Schumacher CM, Senn N, Hasler M, Gschwind S, Hirt AM, Gunther D, Clavien PA, Stark WJ, Beck-Schimmer B. Nanomagnet-based removal of lead and digoxin from living rats. Nanoscale. 2013 Sep 21;5(18):8718-23. doi: 10.1039/c3nr02468g. PMID 23900264